CLINICAL TRIAL: NCT05182593
Title: The Effects of Fermentable Oligosaccharides, Disaccharides, Monosaccharides and Polyols (FODMAPs) in Patients With Irritable Bowel Syndrome
Brief Title: The Effects of FODMAPs in Patients With Irritable Bowel Syndrome
Acronym: Sens-IBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Magnus Simrén, Professor, Sahlgrenska University Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 394-18
Record Dates: First submitted 2021-12-20; First posted 2022-01-10 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Irritable Bowel Syndrome
Keywords: FODMAPs; carbohydrates; gastrointestinal symptoms; IBS
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized, Double-blind, Cross-over Trial
Who Masked: Participant, Investigator
Masking Description: The randomization was done by employees of the hospital that were otherwise not involved in the study by drawing concealed envelops. The interventions were meal boxes which looked similar.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diet 1: moderate/high FODMAP diet. Diet 2: low FODMAP diet. (Experimental): The subjects will follow the moderate/high FODMAP diet as the first intervention, and the low FODMAP diet as the second intervention. The subjects will follow both interventions for seven days.
  Interventions: Other: Diet moderate/high in FODMAPs; Other: Diet low in FODMAPs
- Diet 1: low FODMAP diet. Diet 2: moderate/high FODMAP diet. (Experimental): The subjects will follow the low FODMAP diet as the first intervention, and the moderate/high FODMAP diet as the second intervention. The subjects will follow both interventions for seven days.
  Interventions: Other: Diet moderate/high in FODMAPs; Other: Diet low in FODMAPs

INTERVENTIONS:
Other: Diet moderate/high in FODMAPs — The subjects will obtain meal boxes prepared in the hospital kitchen with a moderately high FODMAP content (23 grams/day)
Other: Diet low in FODMAPs — The subjects will obtain meal boxes prepared in the hospital kitchen with a low FODMAP content (<5 grams/day)

SUMMARY:
Patients with Irritable Bowel Syndrome (IBS) often link their symptoms to foods. Interest in dietary management recently increased, including the use of a low FODMAP diet.

To investigate relation of FODMAPs and IBS, a randomized, double-blind, cross-over trial will be carried out in adult (>18) patients with IBS according to Rome IV criteria. The aim is to assess low FODMAP diet versus moderate/high FODMAP diet in IBS patients.

DETAILED DESCRIPTION:
The study is a randomized, double-blind, cross-over trial.

The aim is to assess the effects of low fermentable oligosaccharides, disaccharides, monosaccharides and polyols (FODMAP) diet compared to moderate/high FODMAP diet in IBS patients on gastrointestinal symptoms and psychological factors. The primary hypothesis is that the low FODMAP diet decreases gastrointestinal symptoms compared to moderate/high FODMAP diet, and that this change is accompanied with reduced psychological distress.

IBS patients (Rome IV) are challenged with FODMAPs in this randomized, double-blinded, cross-over study. The subjects will start with the low FODMAP diet or moderate/high FODMAP diet and cross over to the other intervention (both for 7 days). In between the interventions, there is a wash-out period of at least 14 days. The subjects will receive ready-made meals from the hospital kitchen (lunch and dinner) and in between snacks. The subjects are instructed to buy breakfast themselves and the subjects will receive information on which other foods to avoid, without mentioning 'FODMAPs'. The subjects will follow their usual diet (as before initiation of the study) during the wash-out period.

Primary outcomes are change in gastrointestinal symptoms, assessed by questionnaires, including IBS Severity Scoring System (IBS-SSS) (7-10 day recall and modified daily) and Gastrointestinal Symptom Rating Scale -IBS (GSRS-IBS). A 50-point reduction in IBS-SSS indicates clinical response. Bacterial fermentation (exhaled hydrogen and methane) and visceral sensitivity will be measured using the Lactulose Nutrient Challenge Test. Secondary outcomes are change in psychological factors and assessed by questionnaires, including Central Sensitization Index (CSI), Hospital Anxiety and Depression Scale (HADS), Patient Health Questionnaire (PHQ)-15 and Visceral Sensitivity Index (VSI).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with IBS according to Rome IV criteria

Exclusion Criteria:

* allergy or documented intolerance to food
* severe cardiovascular disease
* severe hepatic disease
* severe neurological disease
* severe psychiatric disease
* celiac disease
* inflammatory bowel diseases
* diabetes
* bowel dysfunction related to previous surgery
* pregnant or lactating women
* use of antibiotics within four weeks before inclusion
* strict avoidance of foods

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Change in Irritable Bowel Syndrome-Severity Scoring System (IBS-SSS) (7-10 days recall questionnaire) | Baseline (day 0), day 7, day 21, day 28
  Irritable Bowel Syndrome-Severity Scoring System (IBS-SSS) is a validated questionnaire that incorporates typical IBS symptoms such as abdominal pain, abdominal distension and bowel dysfunction, as well as quality of life. Subjects rated their symptoms on a visual analogue scale. The maximum achievable score is 500 points (sum of the 5 scales). A reduction in the total IBS-SSS score of at least 50 points is considered to indicate a clinically significant improvement in symptoms. The scale can also be used to classify IBS symptoms severity: <75 points (no symptoms), 75-175 points (mild symptoms), 175-300 points (moderate symptoms) and >300 points (severe symptoms). Measured after both dietary periods and at baseline of both periods.
Change in Irritable Bowel Syndrome-Severity Scoring System (IBS-SSS) (modified, daily IBS-SSS) | Daily during day 7 to 14, and day 21 to 28
  Irritable Bowel Syndrome-Severity Scoring System (IBS-SSS) is a validated questionnaire that incorporates typical IBS symptoms such as abdominal pain, abdominal distension and bowel dysfunction, as well as quality of life. Subjects rated their symptoms on a visual analogue scale. The maximum achievable score is 500 points (sum of the 5 scales). A reduction in the total IBS-SSS score of at least 50 points is considered to indicate a clinically significant improvement in symptoms. The scale can also be used to classify IBS symptoms severity: <75 points (no symptoms), 75-175 points (mild symptoms), 175-300 points (moderate symptoms) and >300 points (severe symptoms). Measured after both dietary periods and at baseline of both periods.
Change in Gastrointestinal Symptom Rating Scale - Irritable Bowel Syndrome (GSRS-IBS) | Baseline (day 0), day 7, day 21, day 28
  Change in Gastrointestinal Symptom Rating Scale - Irritable Bowel Syndrome (GSRS-IBS) measures symptom severity and symptom frequency in IBS patients and is a reliable and validated questionnaire. Thirteen questions are evaluated and rated from 1 (no discomfort at all) to 7 (very severe discomfort) on a Likert scale. The total scores can range from 13 to 91 (sum of the domains). The GSRS-IBS evaluates 5 domains: abdominal pain, bloating, constipation, diarrhea and satiety. Measured after both dietary periods and at baseline of both periods.

SECONDARY OUTCOMES:
Change in stool consistency and frequency, measured by Bristol Stool Form (BSF) | Baseline (day 0), day 7, day 21, day 28
  Change in Bristol Stool Form, stool consistency/frequency per day after both dietary periods
Change in Hospital Anxiety and Depression Scale (HADS) score | Baseline (day 0), day 7, day 21, day 28
  The Hospital Anxiety and Depression Scale (HADS) contains 7 items for depression and 7 for anxiety. Each item is scored from 0 to 3, and therefore the total score per sub-scale can range from 0 to 21. When subjects score >10 on 1 or 2 of the sub-scales, clinically significant psychological distress (anxiety or depression) is likely present. Measured after both dietary periods and at baseline of both periods.
Change in Patient health questionnaire-15 (PHQ-15) | Baseline (day 0), day 7, day 21, day 28
  The (PHQ-15) is a validated questionnaire that evaluates 15 somatic symptoms and can be used as a screening tool for somatization in clinical research. The maximum score for men is 28 and 30 for women due to a question about menstrual problems. Measured after both dietary periods and at baseline of both periods.
Change in Visceral Sensitivity Index (VSI) | Baseline (day 0), day 7, day 21, day 28
  The Visceral Sensitivity Index (VSI) is a validated and reliable psychometric instrument which assesses gastrointestinal symptom-specific anxiety. The VSI contains 15 items that are scored from 0 to 5, therefore the total score can range from 0 to 75. Higher scores indicate more severe gastrointestinal symptom-specific anxiety. Measured after both dietary periods and at baseline of both periods.

OTHER OUTCOMES:
Visceral Sensitivity and Bacterial Fermentation | Baseline (day 0)
  Visceral Sensitivity and Bacterial Fermentation measured by the Lactulose Nutrient Challenge Test. To assess if visceral sensitivity and/or bacterial fermentation are predictors of clinical response to the low FODMAP diet or clinical worsening to the moderate/high FODMAP diet.
Change in microbiota content of frozen fecal samples | Baseline (day 0), day 7, day 21, day 28
  Fecal microbiota analysis using 16 S RNA technique and Dysbiosis Test. Analyses will be done on samples from before and after both dietary periods.
Change in metabolites content | Baseline (day 0), day 7, day 21, day 28
  Frozen urine/serum/fecal samples will be analyzed in the future by gas/liquid chromatography mass spectrometry (metabolomics) analysis.Analyses will be done on samples from before and after both dietary periods.

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Simrén, Professor, Principal Investigator — Göteborg University
Locations (1):
- Magnus Simren, Gothenburg, Non-US/Non-Canadian, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Algera JP, Demir D, Tornblom H, Nybacka S, Simren M, Storsrud S. Low FODMAP diet reduces gastrointestinal symptoms in irritable bowel syndrome and clinical response could be predicted by symptom severity: A randomized crossover trial. Clin Nutr. 2022 Dec;41(12):2792-2800. doi: 10.1016/j.clnu.2022.11.001. Epub 2022 Nov 4. PMID 36384081